CLINICAL TRIAL: NCT00353444
Title: Transcranial Doppler Measurement and Prognosis in Moderate Head Injury
Status: Suspended | Type: Observational
Why Stopped: Technical Conflicts
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Other Study IDs: 27-07TCDHI
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Head Injury
Keywords: head injury; transcranial Doppler; pulsatility index; vasospasm in head injury
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine whether Transcranial Doppler measurements have correlation with neuropsychological test (Galvestone Orientation Amnesia Test), TC image (Marshall Scale) and prognosis (DRS and GOS) in moderate head injury

DETAILED DESCRIPTION:
The head injury is a frequent problem of health, which produces high morbi-mortality. Today is the main cause of death and disability between 18 and 40 years. In addition it originates expensive expenses in health care systems.

Severity of cerebral injury is not only because of impact, it is implicated many physiopathological changes. Decrease or increase of cerebral blood flow (CBF) play important roll formation of edema and intracranial hypertension. Hypoxic/ischemic damage is the final point of both changes.

The transcranial Doppler (TCD) was introduced around 1982. Through TCD can be measured the flow velocity of intracranial arteries, which let us identify changes in diameter in vessels. There are three windows of access to arteries: transtemporal, transorbitary and suboccipital.

The parameter are systolic velocity (S), tele-diastolic velocity (D), mean velocity (M) and pulsatility index (PI). Many studies have been conducted for evaluate utility in head injury, TCD can identify changes that correlate with alteration in CBF intracranial pressure (ICP).

The autoregulatory status is important, TCD with decrement in D and increment in PI could tell us about failure in this issue. An invasive way for estimate cerebral perfusion pressure (CCP) with TCD. The most sensible for fall in is amplitude in FV. However there is more correlation between CPP and PI. Vasospasm can occur post trauma, for identify the Lindegaard ratio (FVcma/FVcia) is useful. The other change, hyperemia, can be demonstrated by continuously increase FV. In post traumatic time is very important identify alterations which could produce ischemia. The measurement of CPP generally is gotten by invasión with ICP determination.

In severe head injury has been demonstrated correlation between ICP and PI, strongest for CPP and PI. Other parameters are oligaemia and vasospasm in the first 24 hours correlate poor outcome.

Because of the non invasive characteristic and good correlation with physiologic and prognosis, we think it is important evaluate if there are a kind of correlation between amnesia and orientation, prognosis and TCD parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman >16 and <50 years with HI less 24 hours in progression and Glasgow between 9 y 12.
2. Man or woman >16 and <50 years with HI and Glasgow l3, with lesions in TC scan.
3. TC scan.
4. Acceptance of family to participate (first grade).

Exclusion Criteria:

1. History of HI with disability
2. History of neurological or psychiatric disease with disability.
3. Existence of systemic injury with life in compromise (massive bleeding, exposition in fracture, hepatic or splenic laceration or in great vessels and shock).
4. Existence of intracranial lesion which needs surgery.
5. Cerebral death certificated by neurologist or neurosurgeon (EEG o arteriography).
6. Management previous in other Hospital.
7. Hemoglobin < 10 g/L

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70
Dates: Start 2006-12; Study Completion 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Torres-Corzo Jaime, Neurosurgeon, Principal Investigator — Hospital Central "Dr. Ignacio Morones Prieto"; Tapia-Perez Humberto, MD, Principal Investigator — Facultad de Medicina UASLP
Locations (1):
- Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí, Mexico